CLINICAL TRIAL: NCT02546427
Title: Phase I Feasibility Study of Accelerated Hypofractionated Whole Pelvic Radiotherapy for Patients With Intermediate-High Risk Prostate Cancer
Brief Title: Hypofractionated Whole Pelvic Radiotherapy of the Prostate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left UCSF and the study was closed without any accruals.
Sponsor: Albert J. Chang (Other)
Responsible Party: Sponsor-Investigator, Albert J. Chang, Assistant Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15551
Record Dates: First submitted 2015-08-27; First posted 2015-09-10 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Step 1: Pelvic Lymph Node Irradiation
  Helical TomoTherapy (HT): 41.25 Gy in 15 fractions of 2.75 Gy each
  Step 2: Treat boost volume to prostate and seminal vesicles
  Acceptable treatment modalities:
  CyberKnife SBRT: 19 Gy in 2 fractions of 9.5 Gy each with SBRT
  Permanent prostate implant (PPI):
  108 Gy for low dose rate PPI with I-125 90 Gy for low dose rate PPI with Pd-103 HDR brachytherapy: 15 Gy in one fraction for HDR
  Interventions: Radiation: Helical TomoTherapy (HT); Radiation: CyberKnife SBRT; Radiation: Permanent Prostate Implant (PPI); Radiation: HDR brachytherapy

INTERVENTIONS:
Radiation: Helical TomoTherapy (HT)
Radiation: CyberKnife SBRT
Radiation: Permanent Prostate Implant (PPI)
Radiation: HDR brachytherapy

SUMMARY:
This is a phase I feasibility study to evaluate the feasibility of hypofractionated whole pelvis radiotherapy in 35 patients with biopsy-proven intermediate- to high-risk prostate cancer as defined by NCCN risk criteria. Patients will have >15% risk of lymph node involvement as defined by the Roach equation 2/3(PSA)+10(Gleason Score-6). Day 0 of the study will be defined as the time of first LHRH/agonist/antagonist injection of hormone therapy. Radiation therapy should begin within 8 weeks (+/- 1 week) after the date of the first LHRH agonist/antagonist injection. Patients will be followed at 6 weeks and then every 3 months for the first 24 months after completion of radiotherapy in a similar schedule to usual standard of care. A history and physical, PSA, testosterone and EPIC-26 questionnaire will be collected at each visit. Any toxicity according to CTCAE v. 4.0 criteria will be documented. An interim analysis for evaluating acute toxicity (≤90 days) will be performed after the first follow-up visit of the20th patient enrolled on protocol. The trial will be terminated if >30% acute grade 2 or >5% grade 3 or greater toxicity is observed as a result of radiation treatment by CTCAE v. 4.0 criteria. Grade 2 toxicity is defined as a minimal, local or noninvasive intervention. Grade 3 toxicity is defined as a severe or medically significant but not immediately life-threatening event requiring hospitalization or prolongation of hospitalization. Previous studies have demonstrated approximately 30% and 5% incidence of Grade 2 and Grade 3 or greater toxicity, respectively, with conventionally fractionated radiotherapy followed by brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intermediate- to high-risk prostate adenocarcinoma (T1c-T3b, PSA >10, and/or Gleason score ≥ 7) who have a greater than 15% risk of lymph node involvement as determined by the Roach equation.
* History/physical examination with digital rectal examination of the prostate within 8 weeks prior to registration
* Zubrod performance status 0-2
* Age ≥18 years
* Ability to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

* Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 5 years.
* Evidence of distant metastases
* Regional lymph node involvement
* Previous radical surgery (prostatectomy) or cryosurgery for prostate cancer
* Previous pelvic irradiation, prostate brachytherapy
* Previous or concurrent cytotoxic chemotherapy for prostate cancer
* Patients with history of inflammatory bowel disease or major bowel surgery.
* Prior transurethral resection of the prostate (TURP) procedure.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Toxicity | 90 days post treatment
  Acute G3 or greater genitourinary or gastrointestinal toxicity as measured by CTCAE v.4

SECONDARY OUTCOMES:
Late Toxicity | From 90 days post treatment until 36 months from start of therapy
  G3 or greater genitourinary or gastrointestinal toxicity as measured by CTCAE v.4
High-Related Quality of Life (HRQOL) | Baseline, week prior to RT, 6 weeks post treatment, and at least every 6 months for the first 2 years.
  EPIC-26 Questionnaire
PSA Complete Response (PSA-CR) | 120-127 days after initiation of therapy
  Via PSA laboratory with PSA level ≤0.3